CLINICAL TRIAL: NCT02408562
Title: A Phase 1, Multicentre, Randomised, Double-blind Study to Assess Safety and Tolerability of Repeated Intracerebroventricular Administration of sNN0031 Infusion Solution to Patients With Parkinson's Disease
Brief Title: Study on Tolerability of Repeat i.c.v. Administration of sNN0031 Infusion Solution in Patients With PD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Issues with development and supply of infusion system for delivery of IMP. Prolonged approval process for the clinical study sNN0031-004.
Sponsor: Newron Sweden AB (Industry)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: sNN0031-004
Record Dates: First submitted 2015-03-05; First posted 2015-04-03 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Becaplermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sNN0031 (Experimental): sNN0031 Infusion Solution (in aCSF) for intracerebroventricular (i.c.v.) administration by an implanted infusion pump
  Interventions: Other: i.c.v. infusion of sNN0031 by an Implanted infusion system
- Placebo (Placebo Comparator): Articifial Cerebro Spinal Fluid (aCSF) for intracerebroventricular (i.c.v.) administration by an implanted infusion pump
  Interventions: Other: i.c.v. infusion of aCSF by an Implanted infusion system

INTERVENTIONS:
Other: i.c.v. infusion of sNN0031 by an Implanted infusion system — I.c.v. infusion during 2 12d cycles separated by 3 mo. 6 mo follow-up after 2nd cycle.
  Other Names: rhPDGF-BB; Medtronic SynchroMed® II Infusion System
  Arms: sNN0031
Other: i.c.v. infusion of aCSF by an Implanted infusion system — I.c.v. infusion during 2 12d cycles separated by 3 mo. 6 mo follow-up after 2nd cycle.
  Other Names: Placebo, Artificial Cerebrospinal fluid; Medtronic SynchroMed® II Infusion System
  Arms: Placebo

SUMMARY:
This is a phase I, randomised, placebo-controlled study to assess the safety and tolerability of two 2-weeks cycles of i.c.v. administration of sNN0031 infusion solution to patients with PD of moderate severity with persisting on-off symptoms in spite of other PD medications.

ELIGIBILITY:
Main Inclusion Criteria:

1. Disease duration ≥ 5 years (diagnosis based on medical history and neurological examination).
2. Male or female, age 30 - 75 years inclusive.
3. Motor fluctuations, with OFF-time >1.5 hours during the day
4. A Hoehn and Yahr stage of 2 to 4 during OFF phase
5. Score >22 on the UPDRS part III during ON phase
6. Patients should be L-dopa responsive and demonstrate at least a 30% decrease in the UPDRS part III score after administration of L-dopa (L-dopa challenge test)
7. Optimised and stable anti-Parkinson treatment for at least 3 months before screening

Main Exclusion Criteria:

1. The patient has any indication of forms of parkinsonism other than idiopathic Parkinson's disease
2. The patient is in a late stage of Parkinson's disease, and is experiencing severe, disabling peak-dose or biphasic dyskinesia and/or unpredictable or widely swinging fluctuations in their symptoms
3. Patients who are on treatment with Duodopa or Apomorphine pump at the time of screening
4. The patient has an implanted shunt for the drainage of CSF or an implanted Central Nervous System (CNS) catheter, or have received neurosurgical intervention related to PD (e.g. deep brain stimulation, thalamotomy etc.) or is scheduled to do so during the trial period
5. Concurrent diagnoses of dementia with a score of 24 or lower on Mini-Mental State Examination (MMSE).
6. The patient is depressed, as indicated by a Hamilton Depression Rating Scale (GRID-HAMD, 17-item scale) score > 17
7. Patients who are at high risk of suicide as judged by the rating of the Columbia Symptoms Suicide Rating Scale (C-SSRS)
8. Patients with a history of increased intracranial pressure
9. Ophthalmologic examination (funduscopy and visual acuity by Early Treatment of Diabetic Retinopathy Study (EDTRS) and perimetry) with clinically significant findings that imply safety concerns for this study
10. The patient has a current clinically significant gastrointestinal, renal, hepatic, endocrine, pulmonary or cardiovascular disease
11. The patient has heart problems or a significant ECG abnormality
12. Uncontrolled hypertension.
13. The patient has in the past experienced psychotic symptoms (e.g. schizophrenia or psychotic depression)
14. The patient has a mental or physical condition which would preclude performing study assessments
15. Alcohol or substance dependence within the prior 12 months, or abuse within 3 months, with the exceptions of nicotine
16. MRI examination with findings of tumours or potential sources of pathological bleedings, or any abnormality that may put the patient at risk
17. History of structural brain disease including tumours and hyperplasia
18. Ongoing or suspected primary or recurrent malignant disease (currently active or in remission for less than one year)
19. Any disorder that precludes a surgical procedure, alters wound healing or renders chronic i.c.v. delivery or device implants medically unsuitable
20. The patient has a history or a current diagnosis of HIV, Hepatitis B or C.
21. Increased susceptibility to infections
22. Women who are pregnant or breast feeding or unwilling to use adequate contraception during the trial (only women of child bearing potential)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Tolerability of sNN0031 [Number of Adverse Events (AE) and Serious Adverse Events (SAE) occurring in each group over the study duration] | 10 months
  Number of AEs and SAEs occurring in each group over the study duration

SECONDARY OUTCOMES:
Peak concentrations of sNN0031 in cerebrospinal fluid during two 14 day continuous infusion cycles | 14 days x 2
  To explore peak concentrations of Platelet Derived Growth Factor-BB (PDGF-BB) levels in cerebrospinal fluid (CSF) during two different treatment cycles of 70 μg sNN0031 each separated by 3 months
Pump flow error rate | 10 months
  Performance of the Medtronic SynchroMed® II Infusion System - Pump flow error rate within 25%
Number of patients with AEs related to the Implanted Infusion System | 10 months
  Number of AEs and SAEs related to the Medtronic SynchroMed® II Infusion System occurring in each group over the study duration

OTHER OUTCOMES:
Explorative evaluation of changes to the Modified Hoehn &Yahr stage following two cycles of sNN0031 | 10 monhts
  To explore the change from baseline in relevant efficacy related variables:
  o Modified Hoehn &Yahr stage
Explorative evaluation of changes to the Unified Parkinson's disease rating scale (UPDRS) following two cycles of sNN0031 | 10 monhts
  To explore the change from baseline in relevant efficacy related variables:
  o Unified Parkinson's disease rating scale (UPDRS)
Explorative evaluation of changes to the Parkinson's disease questionnaire (PDQ-39) following two cycles of sNN0031 | 10 monhts
  To explore the change from baseline in relevant efficacy related variables:
  o Parkinson's disease questionnaire (PDQ-39)
Explorative evaluation of changes to the Dyskinesia rating scale (DRS) following two cycles of sNN0031 | 10 monhts
  To explore the change from baseline in relevant efficacy related variables:
  o Dyskinesia rating scale (DRS)
Explorative evaluation of changes to the o Non-motor symptom scale (NMSS 30) following two cycles of sNN0031 | 10 monhts
  To explore the change from baseline in relevant efficacy related variables:
  o Non-motor symptom scale (NMSS 30)
Changes in presynaptic dopamine transporter (DAT) binding | 10 months
  To explore changes in presynaptic dopamine transporter (DAT) binding in basal ganglia by using DaTscan
Explorative evaluation of potentially relevant biomarkers (inflammatory mediators) in plasma and CSF during and after two cycles of sNN0031 | 10 months
  To explore potentially relevant biomarkers in plasma and CSF - inflammatory mediators.
Explorative evaluation of potentially relevant biomarkers (urate) in plasma and CSF during and after two cycles of sNN0031 | 10 months
  To explore potentially relevant biomarkers in plasma and CSF - urate.
Explorative evaluation of potentially relevant biomarkers (DJ-1/Park7) in plasma and CSF during and after two cycles of sNN0031 | 10 months
  To explore potentially relevant biomarkers in plasma and CSF - DJ-1/Park7.
Explorative evaluation of potentially relevant biomarkers (alpha-synuclein) in plasma and CSF during and after two cycles of sNN0031 | 10 months
  To explore potentially relevant biomarkers in plasma and CSF - alpha-synuclein.
Explorative evaluation of potentially relevant biomarkers (haemoglobin) in plasma and CSF during and after two cycles of sNN0031 | 10 months
  To explore potentially relevant biomarkers in plasma and CSF - haemoglobin.
Explorative evaluation of potentially relevant biomarkers (nitrite/nitrate) in plasma and CSF during and after two cycles of sNN0031 | 10 months
  To explore potentially relevant biomarkers in plasma and CSF - nitrite/nitrate.

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Widner, Prof, Principal Investigator — Lund University Hospital
Locations (5):
- Klinikum-Bremerhaven, Bremerhaven, Germany
- Sweden (2):
  - Lund University Hospital, Lund
  - Karolinska University Hospital Huddinge, Stockholm
- United Kingdom (2):
  - King's College Hospital, London
  - John Radcliffe Hospital, Oxford